CLINICAL TRIAL: NCT05082337
Title: The SAVVY Guidewire in Transcatheter Aortic Valve Replacement Procedures: A Feasibility Study
Brief Title: The SAVVY Guidewire in Transcatheter Aortic Valve Replacement Procedures
Acronym: SAVVY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Collaborators: Institut de Cardiologie de Montréal (Unknown)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, Principal investigator, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRT-2015-02
Record Dates: First submitted 2021-09-21; First posted 2021-10-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Aortic Valve Disease; Transcatheter Aortic Valve Replacement; Aortic Valve Stenosis; Hemodynamic Measurement
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Patient with severe symptomatic aortic stenosis with a clinical indication for TAVR according to the Heart Team criteria will be treated with an approved aortic valve (balloon-expandable or self-expandable aortic valve) and the SAVVY guidewire will be used for the rapid pacing runs and ventricular pressure measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Guidewire (Experimental): The SAVVY guidewire will be used in all TAVR procedures of patients included in the study
  Interventions: Device: SAVVY guidewire

INTERVENTIONS:
Device: SAVVY guidewire — The SAVVY guidewire will be used for rapid pacing runs, valve delivery and for left ventricular pressure measurements pre- and post-THV deployment

SUMMARY:
TAVR patients exhibiting post-procedural residual AR had higher mortality and hospitalization rates due to heart failure, with the extent of this association increasing proportionally to the severity of the regurgitation. Optimizing transcatheter valve performance by intra-procedural hemodynamic evaluation of AR and residual transvalvular gradient remains of high clinical importance.

DETAILED DESCRIPTION:
Continuous technological development and procedural refinements are important to further reduce TAVR peri-procedural complications, facilitate the minimalist strategy and improve clinical outcomes following TAVR. Residual aortic regurgitation (AR) has been one of the main drawbacks of TAVR. TAVR patients exhibiting post-procedural residual AR had higher mortality and hospitalization rates due to heart failure, with the extent of this association increasing proportionally to the severity of the regurgitation.

Various actions could be undertaken to minimize AR and its consequences, either intraprocedural (balloon post-dilation, implantation of a second valve) or during follow-up (diuretic treatment, closest clinical follow-up or percutaneous leakage closure). Thus, an accurate diagnosis of the presence and severity of residual AR post-TAVR is key to implement the proper measures and optimize clinical outcomes.

The use of cardiac imaging remains the gold standard for evaluating AR post-TAVR, limitations of contrast amount along with the subjectivity of AR evaluation by aortic angiography, and the challenges of echocardiography at the time of the TAVR procedure represent a significant drawback. Thus, alternative tools for evaluating the presence and severity of AR would be very helpful in this setting.

Current data supports the implementation of hemodynamic measurements during TAVR procedures in order to improve the clinical decision-making process following valve implantation. However, these actions entail an inherent risk associated with the exchange of catheter-wires. The use of a support guidewire with pressure measurement capabilities would facilitate the hemodynamic evaluation of transcatheter valve performance in a safer and more rapid manner.

The new SAVVY guidewire, with both dedicated pacing properties and allowing a continuous hemodynamic pressure monitoring during the procedure, is a unique system in the field and may represent an important step forward in the process of optimizing the TAVR procedure while facilitating procedural steps.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe symptomatic AS undergoing a TAVR procedure.

Exclusion Criteria:

* Failure to provide signed informed consent.
* Extremely calcified aortic valve (Agatston score >3000 AU)
* Extremely horizontal aorta.
* Severe septal hypertrophy (interventricular septum >15 mm as measured by TTE).
* Extreme tortuosity at the level of the iliofemoral arteries, thoracic or abdominal aorta.
* Prohibitive surgical risk precluding (according to the Heart Team) conversion to open heart surgery in case of a life threatening complication.
* Young patients (<18 Years) and pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Presence of Major complications | Periprocedural
  Presence of major complications related to the SAVVY guidewire including (i) guidewire kink hindering or preventing the advancement of the transcatheter valve system
Presence of Major vascular complications | Periprocedural
  Major vascular complications related to the SAVVY guidewire are defined as stroke, bleeding or left ventricular perforation
Number of transcatheter valve malpositioning | Periprocedural
  Pacing capture failure translating into valve malpositioning. Valve malpositiong will be evaluated by a landing site to low or too high, leading to hemodynamically unfavorable results.
Number of valve embolization | Periprocedural
  Pacing capture failure translating into valve embolization
Number of effective rapid pacing run | Periprocedural
  Effective rapid pacing will be defined as an adequate ventricular pacing capture for a minimum of 10 seconds, with no capture loss, and leading to a reduction of aortic pressure of at least 50%, with/or a systolic pressure value <60 mmHg. Efficacy will be assessed by the physician.
Number of accurate ventricular pressure | Periprocedural
  Accurate ventricular pressure will be defines as a pressure wire measurements similar (differences <5 mmHg) to those obtained simultaneously with a pigtail catheter in the same cavity or vascular segment (differences <5 mmHg in SBP, differences <5 mmHg in LVEDP).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - ICM, Montreal, Quebec
  - IUCPQ, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Fleisher LA, Jneid H, Mack MJ, McLeod CJ, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A. 2017 AHA/ACC Focused Update of the 2014 AHA/ACC Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2017 Jun 20;135(25):e1159-e1195. doi: 10.1161/CIR.0000000000000503. Epub 2017 Mar 15. No abstract available. PMID 28298458
- [Background] Popma JJ, Deeb GM, Yakubov SJ, Mumtaz M, Gada H, O'Hair D, Bajwa T, Heiser JC, Merhi W, Kleiman NS, Askew J, Sorajja P, Rovin J, Chetcuti SJ, Adams DH, Teirstein PS, Zorn GL 3rd, Forrest JK, Tchetche D, Resar J, Walton A, Piazza N, Ramlawi B, Robinson N, Petrossian G, Gleason TG, Oh JK, Boulware MJ, Qiao H, Mugglin AS, Reardon MJ; Evolut Low Risk Trial Investigators. Transcatheter Aortic-Valve Replacement with a Self-Expanding Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1706-1715. doi: 10.1056/NEJMoa1816885. Epub 2019 Mar 16. PMID 30883053
- [Background] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Background] Genereux P, Head SJ, Hahn R, Daneault B, Kodali S, Williams MR, van Mieghem NM, Alu MC, Serruys PW, Kappetein AP, Leon MB. Paravalvular leak after transcatheter aortic valve replacement: the new Achilles' heel? A comprehensive review of the literature. J Am Coll Cardiol. 2013 Mar 19;61(11):1125-36. doi: 10.1016/j.jacc.2012.08.1039. Epub 2013 Jan 30. PMID 23375925
- [Background] Athappan G, Patvardhan E, Tuzcu EM, Svensson LG, Lemos PA, Fraccaro C, Tarantini G, Sinning JM, Nickenig G, Capodanno D, Tamburino C, Latib A, Colombo A, Kapadia SR. Incidence, predictors, and outcomes of aortic regurgitation after transcatheter aortic valve replacement: meta-analysis and systematic review of literature. J Am Coll Cardiol. 2013 Apr 16;61(15):1585-95. doi: 10.1016/j.jacc.2013.01.047. PMID 23500308
- [Background] Nishimura RA, Carabello BA. Hemodynamics in the cardiac catheterization laboratory of the 21st century. Circulation. 2012 May 1;125(17):2138-50. doi: 10.1161/CIRCULATIONAHA.111.060319. No abstract available. PMID 22547754
- [Background] Pibarot P, Hahn RT, Weissman NJ, Monaghan MJ. Assessment of paravalvular regurgitation following TAVR: a proposal of unifying grading scheme. JACC Cardiovasc Imaging. 2015 Mar;8(3):340-360. doi: 10.1016/j.jcmg.2015.01.008. PMID 25772838
- [Background] Liao YB, Deng XX, Meng Y, Zhao ZG, Xiong TY, Meng XJ, Zuo ZL, Li YJ, Cao JY, Xu YN, Chen M, Feng Y. Predictors and outcome of acute kidney injury after transcatheter aortic valve implantation: a systematic review and meta-analysis. EuroIntervention. 2017 Apr 20;12(17):2067-2074. doi: 10.4244/EIJ-D-15-00254. PMID 27890858
- [Background] Kamioka N, Wells J, Keegan P, Lerakis S, Binongo J, Corrigan F, Condado J, Patel A, Forcillo J, Ogburn L, Dong A, Caughron H, Simone A, Leshnower B, Devireddy C, Mavromatis K, Guyton R, Stewart J, Thourani V, Block PC, Babaliaros V. Predictors and Clinical Outcomes of Next-Day Discharge After Minimalist Transfemoral Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2018 Jan 22;11(2):107-115. doi: 10.1016/j.jcin.2017.10.021. PMID 29348004